CLINICAL TRIAL: NCT00465504
Title: Comparison of Iontophoresis of Lidocaine and Eutectic Mixture of Local Anesthetics (EMLA®) Cream Versus Subcutaneous Injections of Lidocaine and EMLA® for Pain Relief in Intra-articular Corticosteroid Injections in Children With Juvenile Idiopathic Arthritis: A Randomized Clinical Trial
Brief Title: Comparison of Two Different Methods of Delivering Local Analgesia During Intra-articular Corticosteroid Injections in Children With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Childrens Hospital Foundation (Other)
Responsible Party: Dr. Peter Malleson, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H06-70290
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Pain
Keywords: local analgesia; intra-articular corticosteroid injection; iontophoresis; Local analgesia for intra-articular corticosteroid injection
MeSH Terms: conditions — Pain | interventions — Iontophoresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: iontophoresis — See Detailed Description.

SUMMARY:
Chronic arthritis (inflammation of joints) in children is known as Juvenile Idiopathic Arthritis (JIA). Often, to control the swelling and to help reduce the pain in the joint, medications (steroids) are injected into the joint. These injections are sometimes painful, even if we use local anesthetics (lidocaine) to numb the skin; in fact, lidocaine injection is often the most painful part of the procedure. There is an alternate method called iontophoresis that uses an electric current to push lidocaine into the skin and deeper tissues avoiding the anesthetic injection. Very little work has been done to see if this is actually an effective way of numbing the skin in children having painful procedures such as joint injections. In this study, we will compare two groups of children with JIA having steroid injections into their joints: one group will get lidocaine by iontophoresis and the other will get it by the usual injection method. We will assess the child's pain during the steroid injection and compare the two groups to see if children who are given local anesthetic by iontophoresis experience less pain. The results of this study will provide new information about the effectiveness of the iontophoresis method, and whether or not this would be a better way to give local anesthetic for children undergoing other kinds of painful procedures.

DETAILED DESCRIPTION:
Research method: This study will be a prospective, randomized clinical trial comparing two methods of delivery of local anesthesia for intra-articular corticosteroids injection (IACI) in children with JIA. There will be two study groups:

1. Children receiving analgesia with subcutaneous lidocaine 2% and EMLA® cream (Rheumatology Division standard of care arm) (n=33)
2. Children receiving analgesia with iontophoresis and EMLA® cream (experimental arm) (n=33).

About one child with JIA per week receives IACI in our institution. To minimize procedural variations in this study, we will select children undergoing knee (by far the most commonly injected joint) IACI by the Pediatric Rheumatology service at BC Children's Hospital. Randomization will be achieved with a Microsoft Access 2003 program. Our primary outcome measures will be change in pain between baseline pain assessed immediately prior to the corticosteroid injection, immediately after the local anesthetic application, and after the corticosteroid injection, using a 10-cm visual analogue scale (VAS, a continuous variable) and the Facial Pain Scale-Revised (FPS-R) scores (a categorical variable). The change in pain will be analyzed using Student's t-test for VAS scores and with Mann-Whitney U test for FPS-R scores. Descriptive statistics for demographic and auxiliary clinical variables will be presented in tables, including mean, range and standard deviation for continuous variables and median, range and percentiles for categorical variables.

Adverse events from EMLA® or iontophoresis will also be recorded (i.e. tingling, redness, blanching, itching, blistering, or pain). Data collected will consist of the child's age, gender, JIA type and duration, number and sites of previous IACIs, and other medications used and will have no patient identifiers (such as name, date of birth, personal health number).

ELIGIBILITY:
Inclusion Criteria:

* All children aged >4 years with JIA and active arthritis of at least one knee despite treatment with NSAIDs or disease modifying anti-rheumatic drugs who are undergoing an IACI will be eligible.

Exclusion Criteria:

* Children who are allergic to lidocaine, any ingredient used in EMLA® cream or the iontophoresis pads
* Have electrically-sensitive support systems (i.e. pacemakers)
* Damaged skin or signs of infection at the injection site
* Suffering from a coagulation disorder
* Unable to evaluate pain

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The main outcome measure will be the change in level of pain, from baseline pain at maximal range of motion (ROM) to pain associated with the procedure, as rated by the child and parent. This approach contrasts with measurement of absolute levels of pain

SECONDARY OUTCOMES:
Secondary outcomes will include pain scores during the procedure as follows: 1 during the application of the analgesic agents and 2. at a 24 hours follow-up telephone call. Will be attained by July 2008.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Malleson, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada